CLINICAL TRIAL: NCT02257060
Title: Evaluation of a Multi-Electrode Linear Type Ablation Catheter for Endocardial Ablation of Patients With Right Atrial Flutter
Brief Title: LINEAR II - LME-159 Evaluation of a Multi-Electrode Linear Type Ablation Catheter
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LINEAR II
Record Dates: First submitted 2014-09-02; First posted 2014-10-06 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cavotricuspid Isthmus Dependent Right Atrial Flutter
Keywords: Endocardial Ablation; Atrial Flutter; Cavotricuspid Isthmus
MeSH Terms: conditions — Atrial Flutter

ARMS (1):
- Endocardial Ablation (Experimental)
  Interventions: Procedure: Endocardial Ablation

INTERVENTIONS:
Procedure: Endocardial Ablation
  Other Names: Radiofrequency (RF) ablation with the; - Linear Type Ablation Catheter; - nMARQ™ Multi-Channel RF Generator with Software V2.4.0; - Linear Ablation Connection Cable

SUMMARY:
The Linear II study is a prospective, single center, non-randomized, interventional feasibility study with the purpose of assessing acute safety of the Multi-Electrode Linear Type Ablation Catheter and the performance of the product when used for the treatment of symptomatic CTI (cavotricuspid isthmus) dependent right atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

* At least one symptomatic episode of typical CTI dependent right atrial flutter documented by 12 lead ECG, Holter monitor, transtelephonic event monitor, telemetry strip, or implanted device.
* Age 18 years or older.

Exclusion Criteria:

* Previous typical CTI dependent right atrial flutter ablation
* Uncontrolled heart failure or NYHA function class IV
* MI within the past 2 months
* Any cardiac surgery (i.e. CABG) within the past 2 months
* Subjects that have ever undergone valvular cardiac surgical procedure (ie, ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve)
* Awaiting cardiac transplantation or other cardiac surgery within the next 6 months
* Documented thromboembolic event (including TIA) within the past 12 months
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
* Active illness or active systemic infection or sepsis
* Unstable angina
* History of blood clotting or bleeding abnormalities
* Contraindication to anticoagulation (eg, heparin or warfarin)
* Life expectancy less than 6 months
* Presence of intracardiac thrombus, myxoma, interatrial baffle or patch, tumor or other abnormality that precludes catheter introduction or manipulation
* Presence of a condition that precludes vascular access
* Women of child bearing potential whom are pregnant, lactating, or planning to become pregnant during the course of the clinical investigation
* Currently enrolled in another device, biologics, or drug study
* Contraindication for use of the investigational catheter, as indicated in the respective Instructions For Use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety | 7 Days
  Incidence of early onset (within 7 days of ablation procedure) primary AEs
Acute performance | This outcome measure will be assessed during the procedure but after 30 minutes (or more) of the initial ablation
  Acute procedural success as confirmed complete bidirectional conduction block across the CTI (assess ≥30 min following last RF application)

SECONDARY OUTCOMES:
Safety | Until one-month follow-up
  Incidence of Serious Adverse Events during follow-up
Acute Efficacy | Within 30 Days
  Right atrial flutter recurrence within 30 days
Procedural data | During Procedure
  Ablation parameters, including:
  * Total RF ablation time
  * Temperature
  * Contact Force Procedural time Total fluoroscopy time

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Grimaldi, Principal Investigator — Miulli Hospital